CLINICAL TRIAL: NCT06979609
Title: Secondary Prophylaxis of Recurrent Clostridioides Difficile Infections During Systemic Antibiotics With Vancomycin: A Randomized Controlled Trial
Brief Title: Secondary Prevention of Clostridioides Difficile Using Vancomycin
Acronym: SPORES-V
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Emily McDonald, Associate Professor of General Internal Medicine, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2025-11089
Record Dates: First submitted 2025-05-13; First posted 2025-05-20 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Clostridioides Difficile Infection; Clostridioides Difficile Infection Recurrence; Clostridoides Difficile Associated Disease
Keywords: Clostridioides difficile; Clostridium difficile; Vancomycin; Prophylaxis; C. difficile; Recurrence; CDI
MeSH Terms: conditions — Clostridium Infections; Recurrence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Vancomycin Prophylaxis (Experimental): Vancomycin 125mg PO BID for the duration of antibiotic re-exposure + 125mg PO QD for 7 days
  Interventions: Drug: Oral Vancomycin Prophylaxis
- Placebo (Placebo Comparator): 2 capsules PO BID for the duration of antibiotic re-exposure + 1 capsule PO QD for 7 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral Vancomycin Prophylaxis — 125mg PO BID for the duration of antibiotic re-exposure + 125mg PO QD for 7 days
  Arms: Oral Vancomycin Prophylaxis
Drug: Placebo — 2 capsules PO BID for the duration of antibiotic re-exposure + 1 capsule PO QD x 7 days
  Arms: Placebo

SUMMARY:
Re-exposure to systemic antibiotics (i.e., antibiotics absorbed into the bloodstream) is common after a Clostridioides difficile infection (CDI) and is the strongest risk factor for a recurrent episode. Oral vancomycin to prevent a recurrence during antibiotic re-exposure may reduce this risk but the data supporting this practice are limited. The aim of this trial is:

1) Does oral vancomycin prophylaxis prevent CDI recurrences in patients with recent CDI (within 120 days) and who are re-exposed to systemic antibiotics?

The trial will compare oral vancomycin to placebo.

Participants will:

* Take the study drug (either vancomycin or placebo) twice daily for the duration of systemic antibiotics plus once daily for 7 days after completion of systemic antibiotics.
* Attend an in-person follow-up at day 56
* Respond to weekly electronic questionnaires

DETAILED DESCRIPTION:
Clostridioides difficile is a gram-positive spore-forming anaerobic bacteria that can cause severe diarrhea through colitis. While the incidence of CDI is decreasing in Canada it remains a major cause of nosocomial infections. The annual incidence of CDI in Canada is 16,000 cases with 1,300 (8.1%) associated deaths. Estimates suggest that CDI is associated with annual economic losses of ~$150 million in Canada and that 23% of these losses are attributable to recurrent cases.

Despite appropriate treatment, approximately 20% of CDI cases experience a recurrence. Recurrent CDI (rCDI) is associated with a higher risk of death than index episodes. Although treatments such as fidaxomicin reduce the recurrence rate of CDI by approximately ~10%, cost and availability prohibit their widespread use and a substantial risk of recurrence remains (10-15%). Thus, rCDI is associated with significant morbidity, mortality, and economic cost, and consequently prevention is a substantially unmet clinical need.

Antibiotic re-exposure following completion of CDI treatment is common and is one of the strongest risk factors for CDI recurrence. In a study of 18,246 index cases of CDI, 7,730 were re-exposed to antibiotics within 8 weeks of completion of CDI treatment. Antibiotic re-exposure was the strongest predictor of rCDI with an adjusted odds ratio of 3.2 (95% Confidence Interval [95%CI]=2.9-3.4). Although avoidance of antibiotics after an index episode of CDI would be an ideal prevention strategy, it is frequently unavoidable. Therefore, strategies to reduce the recurrence rate of CDI arising from antibiotic re-exposure are of significant clinical interest.

The pathogenesis of rCDI is thought to involve persistent C. difficile colonization in a patient with an already vulnerable microbiome that is further disrupted by re-exposure to antibiotics. Vancomycin prophylaxis has been proposed as a potential strategy to reduce the risk of rCDI by inhibiting the proliferation of C. difficile during antibiotic re-exposure.

Observational evidence suggests that vancomycin prophylaxis may reduce the recurrence rate of CDI. In a Canadian study of 551 episodes of CDI with antibiotic re-exposure, patients who received vancomycin prophylaxis (n=227, 41.2%) experienced significantly less rCDI after adjusting for age (adjusted hazard ratio=0.59, 95% CI=0.43-0.80). This benefit was only identified following recurrent episodes of CDI. However, the evidence base is inconsistent, as another study found a benefit only in patients with a first episode of CDI and another suggested no benefit at all. These inconsistencies could be attributable to varying degrees of confounding by indication, ascertainment bias, immortal time bias, and a competing risk of mortality, which preclude firm conclusions from observational studies.

A single randomized controlled trial (RCT) of primary oral vancomycin prophylaxis in patients at high risk of CDI and who continued to receive systemic antibiotics demonstrated benefit in the prevention of healthcare-onset CDI (placebo 6/50 [12.0%] versus prophylaxis 0/50 [0%], P=0.03). Results of this trial are limited by its open-label design which may have led to ascertainment bias and an extremely high loss to follow-up (>50%) for the overall rCDI outcome. No RCTs of vancomycin prophylaxis for the prevention of rCDI during antibiotic re-exposure have been published to date. There is one small RCT of vancomycin prophylaxis versus placebo, randomized in a 2:1 ratio, underway with a target enrollment of 108 participants. This RCT uses a 10-day fixed duration of oral vancomycin; however, observational evidence suggests that vancomycin prophylaxis is more effective when given for ≥50% of the duration of systemic antibiotics. Thus, if the trial is negative, dosing based on the duration of antibiotic re-exposure might prove effective. Further, while this trial is appreciated, it is underpowered and unlikely to provide definitive evidence regardless of the result.

Guidelines are heterogeneous in their recommendations for vancomycin prophylaxis following antibiotic re-exposure. Whereas the American College of Gastroenterology and AMMI Canada recommend consideration of prophylaxis, the Infectious Disease Society of America refrain from making a recommendation, and the European Society of Clinical Microbiology and Infectious Diseases discourage prophylaxis. Heterogeneous conclusions from observational studies and conflicting international guideline recommendations implies clinical equipoise. Therefore, to definitively determine whether vancomycin prophylaxis is an efficacious strategy to prevent rCDI during antibiotic re-exposure, the investigators propose a randomized double-blind trial comparing vancomycin prophylaxis to placebo for patients with CDI in the past 120 days who are re-exposed to antibiotics. The proposed trial will directly inform clinical practice on the use of vancomycin for CDI prophylaxis during antibiotic re-exposure. The results are expected to be of international importance given the high incidence and economic burden of rCDI and because oral vancomycin is inexpensive, safe, and widely accessible.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient or outpatient adults (≥18 years old) treated at the participating institutions.
* An episode of CDI within the preceding 120 days (rationale in 2.4), diagnosed by both a positive C. difficile assay (including PCR toxin gene detection47, toxin enzyme immunoassay, and/or cell cytotoxicity neutralization assay29) and the presence of either ≥3 unformed stools in <24 hours with a duration >24 hours, endoscopic/histologic evidence of pseudomembranous colitis, or ileus29.
* Treatment of the qualifying CDI episode with vancomycin or fidaxomicin for ≥10 days, clinical cure (≤3 unformed stool per 24 hours in ≥2 days10) by the conclusion of therapy, and ≥1 day has elapsed since cessation of CDI treatment.
* Receipt of ≤3 days of at least one oral or intravenous systemic antibiotic for the treatment of an intercurrent confirmed or suspected bacterial infection, for which therapy is planned for at least one additional consecutive day in duration.

Exclusion Criteria:

* Treatment of the qualifying episode of CDI with metronidazole monotherapy or intravenous immunoglobulins.
* Planned treatment with or treatment of the qualifying episode of CDI with fecal microbiota transplantation (FMT), bezlotoxumab, VOWST, or REBYOTA.
* Inability to take medications orally or crushed by nasogastric tube.
* Prior total colectomy.
* Severe intolerance or allergy to oral vancomycin.
* Lack of achievement of clinical cure during the treatment of the qualifying CDI episode
* Ongoing or <1 day since receiving CDI treatment or ongoing or <1 days since receipt of CDI-active antibiotics, including oral vancomycin, oral or intravenous metronidazole, or fidaxomicin.
* The qualifying antibiotic is solely for prophylaxis (e.g., once daily trimethoprim sulfamethoxazole) or the patient is anticipated to require systemic antibiotics for >4 weeks (e.g., lifelong suppressive therapy or for the treatment of left-sided endocarditis or a deep-seated abscess).
* Patients on ongoing systemic antibiotics since the completion of treatment for the qualifying episode of CDI that have not been interrupted by at least one day.
* Patients admitted to a palliative care ward or is anticipated to die within 3 months of enrollment from another illness.
* The qualifying antibiotic is non-systemic or is not considered a significant risk factor for CDI including: topical antibiotics, azithromycin, clarithromycin, nitrofurantoin, intravenous vancomycin, minocycline, tetracycline, doxycycline, and oral fosfomycin.
* Prior enrollment in this trial.
* Inability to consent without a healthcare proxy.
* Lack of health insurance.
* Anticipated transfer to a site not involved in this trial or to a palliative care ward.
* Patient declared anticipated inability to participate in study follow-up or lack of means for contact in the outpatient setting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
CDI Recurrence | 56 Days
  Patients reporting diarrhea will be brought in for an in-person appointment that is standard of care for patients with potential rCDI and investigated as appropriate clinically without unblinding. Additionally, patients and/or their proxy will be instructed to contact the study team if they believe they are having a recurrence between contacts. Patients will be able to come be assessed for potential recurrence by infectious diseases physicians at each site (who may or may not be a part of the study) or could see their usual doctors. Recurrence will be assessed by clinical record review (chart, laboratory, pharmacy records) and any direct patient interview.
  CDI recurrence will be defined by 1) three or more unformed stools in a 24-hour period, 2) a positive PCR for toxin gene or and/or detection of toxin by enzyme immunoassay or cell cytotoxicity neutralization assay, and 3) administration of CDI treatment. This is similar to the definition used in the NEJM fidaxomicin trial.

SECONDARY OUTCOMES:
Late CDI Recurrence | 90 Days
  As per the primary outcome.
All-Cause Mortality | 90 Days
  Patients present for their day 56 in-person follow-up are considered alive. Those responding to weekly/bi-weekly surveys (text/email/phone) are considered alive at the response time. If a patient misses the day 56 follow-up, the investigators will review their hospital file for death. If unclear, the investigators will contact the patient or proxy by phone. If unreachable and unresponsive to surveys, the investigators will check obituaries.
  After day 56, survey responses confirm vital status. If there is no response to the day 90 survey by day 95, the investigators will review the hospital file, check obituaries, and then attempt phone contact with the patient or proxy. If unsuccessful, the investigators will send a registered letter. Without a response, the patient will be recorded as lost to follow-up.
Discontinuation of the Study Drug Due to Adverse Event | 56 Days
  During the in-person visit on Day 56 the investigators will inquire about adherence to the study drug and completion of the prescribed course. If the course was not completed, the investigators will inquire as to the reason why. Patients reporting cessation of the study drug due to an adverse event will be recorded as such.
Emergency Room Visits or Hospital Admissions | 90 Days
  Within 90 days the investigators will look in the chart and the patient email/text surveys for the first episode of each of emergency room visit and/or hospital admission and record the date. Patient charts will also be flagged for immediate review should they visit the emergency room or be admitted to study centres. With explicit written patient consent, medical records from outside hospitals will be also requested for review if they report presenting elsewhere.

CONTACTS AND LOCATIONS:
Overall Officials: Todd C. Lee, MD MPH, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Connor J. Prosty, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Prehn J, Reigadas E, Vogelzang EH, Bouza E, Hristea A, Guery B, Krutova M, Noren T, Allerberger F, Coia JE, Goorhuis A, van Rossen TM, Ooijevaar RE, Burns K, Scharvik Olesen BR, Tschudin-Sutter S, Wilcox MH, Vehreschild MJGT, Fitzpatrick F, Kuijper EJ; Guideline Committee of the European Study Group on Clostridioides difficile. European Society of Clinical Microbiology and Infectious Diseases: 2021 update on the treatment guidance document for Clostridioides difficile infection in adults. Clin Microbiol Infect. 2021 Dec;27 Suppl 2:S1-S21. doi: 10.1016/j.cmi.2021.09.038. Epub 2021 Oct 20. PMID 34678515
- [Background] Johnson S, Lavergne V, Skinner AM, Gonzales-Luna AJ, Garey KW, Kelly CP, Wilcox MH. Clinical Practice Guideline by the Infectious Diseases Society of America (IDSA) and Society for Healthcare Epidemiology of America (SHEA): 2021 Focused Update Guidelines on Management of Clostridioides difficile Infection in Adults. Clin Infect Dis. 2021 Sep 7;73(5):e1029-e1044. doi: 10.1093/cid/ciab549. PMID 34164674
- [Background] McDonald LC, Gerding DN, Johnson S, Bakken JS, Carroll KC, Coffin SE, Dubberke ER, Garey KW, Gould CV, Kelly C, Loo V, Shaklee Sammons J, Sandora TJ, Wilcox MH. Clinical Practice Guidelines for Clostridium difficile Infection in Adults and Children: 2017 Update by the Infectious Diseases Society of America (IDSA) and Society for Healthcare Epidemiology of America (SHEA). Clin Infect Dis. 2018 Mar 19;66(7):987-994. doi: 10.1093/cid/ciy149. PMID 29562266
- [Background] Kelly CR, Fischer M, Allegretti JR, LaPlante K, Stewart DB, Limketkai BN, Stollman NH. ACG Clinical Guidelines: Prevention, Diagnosis, and Treatment of Clostridioides difficile Infections. Am J Gastroenterol. 2021 Jun 1;116(6):1124-1147. doi: 10.14309/ajg.0000000000001278. PMID 34003176
- [Background] San-Juan R, Origuen J, Campion K, Fernandez-Ruiz M, Diaz-Pollan B, Callejas-Diaz A, Candela G, Orellana MA, Lora D, Llorente Munoz I, Garcia MT, Martinez-Una M, Ferrari JM, Aguado JM. Evaluation of the effectiveness and safety of oral vancomycin versus placebo in the prevention of recurrence of Clostridioides difficile infection in patients under systemic antibiotic therapy: a phase III, randomised, double-blind clinical trial. BMJ Open. 2023 Sep 13;13(9):e072121. doi: 10.1136/bmjopen-2023-072121. PMID 37709311
- [Background] Maraolo AE, Mazzitelli M, Zappulo E, Scotto R, Granata G, Andini R, Durante-Mangoni E, Petrosillo N, Gentile I. Oral Vancomycin Prophylaxis for Primary and Secondary Prevention of Clostridioides difficile Infection in Patients Treated with Systemic Antibiotic Therapy: A Systematic Review, Meta-Analysis and Trial Sequential Analysis. Antibiotics (Basel). 2022 Jan 30;11(2):183. doi: 10.3390/antibiotics11020183. PMID 35203786
- [Background] Johnson SW, Brown SV, Priest DH. Effectiveness of Oral Vancomycin for Prevention of Healthcare Facility-Onset Clostridioides difficile Infection in Targeted Patients During Systemic Antibiotic Exposure. Clin Infect Dis. 2020 Aug 22;71(5):1133-1139. doi: 10.1093/cid/ciz966. PMID 31560051
- [Background] McDonald EG, Prosty C, Hanula R, Bortolussi-Courval E, Albuquerque AM, Tong SYC, Hamilton F, Lee TC. Observational versus randomized controlled trials to inform antibiotic treatment durations: a narrative review. Clin Microbiol Infect. 2023 Feb;29(2):165-170. doi: 10.1016/j.cmi.2022.09.002. Epub 2022 Sep 13. PMID 36108947
- [Background] Connor KA, Conn KM. Analysis of the impact of secondary prophylaxis on Clostridioides difficile recurrence in critically ill adults. SAGE Open Med. 2020 Jun 12;8:2050312120930898. doi: 10.1177/2050312120930898. eCollection 2020. PMID 32587690
- [Background] Caroff DA, Menchaca JT, Zhang Z, Rhee C, Calderwood MS, Kubiak DW, Yokoe DS, Klompas M. Oral vancomycin prophylaxis during systemic antibiotic exposure to prevent Clostridiodes difficile infection relapses. Infect Control Hosp Epidemiol. 2019 Jun;40(6):662-667. doi: 10.1017/ice.2019.88. Epub 2019 Apr 29. PMID 31030679
- [Background] Najjar-Debbiny R, Barnett-Griness O, Arbel A, Cohen S, Weber G, Amar M, Yassin R, Greenfeld I, Shehadeh S, Saliba W. Secondary prophylaxis for Clostridioides difficile infection for patients on non-C. difficile antibiotics: a retrospective cohort study. Microbes Infect. 2024 Jul-Aug;26(5-6):105349. doi: 10.1016/j.micinf.2024.105349. Epub 2024 May 6. PMID 38719086
- [Background] Van Hise NW, Bryant AM, Hennessey EK, Crannage AJ, Khoury JA, Manian FA. Efficacy of Oral Vancomycin in Preventing Recurrent Clostridium difficile Infection in Patients Treated With Systemic Antimicrobial Agents. Clin Infect Dis. 2016 Sep 1;63(5):651-3. doi: 10.1093/cid/ciw401. Epub 2016 Jun 17. PMID 27318333
- [Background] Carignan A, Poulin S, Martin P, Labbe AC, Valiquette L, Al-Bachari H, Montpetit LP, Pepin J. Efficacy of Secondary Prophylaxis With Vancomycin for Preventing Recurrent Clostridium difficile Infections. Am J Gastroenterol. 2016 Dec;111(12):1834-1840. doi: 10.1038/ajg.2016.417. Epub 2016 Sep 13. PMID 27619835
- [Background] Abujamel T, Cadnum JL, Jury LA, Sunkesula VC, Kundrapu S, Jump RL, Stintzi AC, Donskey CJ. Defining the vulnerable period for re-establishment of Clostridium difficile colonization after treatment of C. difficile infection with oral vancomycin or metronidazole. PLoS One. 2013 Oct 2;8(10):e76269. doi: 10.1371/journal.pone.0076269. eCollection 2013. PMID 24098459
- [Background] Seekatz AM, Rao K, Santhosh K, Young VB. Dynamics of the fecal microbiome in patients with recurrent and nonrecurrent Clostridium difficile infection. Genome Med. 2016 Apr 27;8(1):47. doi: 10.1186/s13073-016-0298-8. PMID 27121861
- [Background] Sethi AK, Al-Nassir WN, Nerandzic MM, Bobulsky GS, Donskey CJ. Persistence of skin contamination and environmental shedding of Clostridium difficile during and after treatment of C. difficile infection. Infect Control Hosp Epidemiol. 2010 Jan;31(1):21-7. doi: 10.1086/649016. PMID 19929371
- [Background] Kimura T, Snijder R, Sugitani T. Characterization and risk factors for recurrence of Clostridioides (Clostridium) difficile infection in Japan: A nationwide real-world analysis using a large hospital-based administrative dataset. J Infect Chemother. 2019 Aug;25(8):615-620. doi: 10.1016/j.jiac.2019.03.011. Epub 2019 Apr 12. PMID 30987950
- [Background] Zilberberg MD, Reske K, Olsen M, Yan Y, Dubberke ER. Risk factors for recurrent Clostridium difficile infection (CDI) hospitalization among hospitalized patients with an initial CDI episode: a retrospective cohort study. BMC Infect Dis. 2014 Jun 4;14:306. doi: 10.1186/1471-2334-14-306. PMID 24898123
- [Background] Deshpande A, Pasupuleti V, Thota P, Pant C, Rolston DD, Hernandez AV, Donskey CJ, Fraser TG. Risk factors for recurrent Clostridium difficile infection: a systematic review and meta-analysis. Infect Control Hosp Epidemiol. 2015 Apr;36(4):452-60. doi: 10.1017/ice.2014.88. Epub 2015 Jan 28. PMID 25626326